CLINICAL TRIAL: NCT00709345
Title: Effectiveness of a Cognitive Behavioral Treatment for Reducing Atypical Antipsychotic Medication Health Risks in People With Serious Mental Illness
Brief Title: Behavioral Intervention to Reduce Novel Antipsychotic Medication Health Risks
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jeffrey Kelly, Professor of Psychiatry and Behavioral Medicine, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH078576 (NIH); R01MH078576 (NIH)
Record Dates: First submitted 2008-06-30; First posted 2008-07-03 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Mental Illness
Keywords: Antipsychotic Medications; Behavioral Interventions
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Home (Experimental): Participants will receive cognitive behavioral sessions.
  Interventions: Behavioral: Cognitive behavioral sessions
- Control (Active Comparator): Participants will receive time-matched attention control sessions.
  Interventions: Behavioral: Time-matched attention control sessions

INTERVENTIONS:
Behavioral: Cognitive behavioral sessions — Participants will receive 26 weekly 1-hour small-group sessions and 26 weekly 30-minute individual sessions with a study facilitator. After completing treatment, participants will also receive 6 monthly 1-hour booster sessions. All sessions will focus on promoting healthy behaviors, dieting, and exercise.
  Arms: Group Home
Behavioral: Time-matched attention control sessions — Participants will receive 26 weekly 1-hour small-group sessions and 26 weekly 30-minute individual sessions with a study facilitator. After completing treatment, participants will also receive 6 monthly 1-hour booster sessions. All sessions will focus on improving communications, developing healthy techniques for coping with stress, and resolving conflicts.
  Arms: Control

SUMMARY:
This study will evaluate the effectiveness of a cognitive behavioral treatment in reducing significant medical risk factors often associated with people who have a serious mental illness and are taking atypical antipsychotic medications.

DETAILED DESCRIPTION:
Serious mental illness encompasses a large range of symptoms varying in severity, but generally includes symptoms described as both positive and negative. Positive symptoms include confused thinking, delusions, and hallucinations, while negative symptoms include lack of emotion and depression. Because novel or atypical antipsychotic medications target both positive and negative symptoms and have fewer side effects than other medications, they make up the current standard of care for the treatment of many mental illnesses. However, there is growing concern that the psychiatric benefits associated with atypical antipsychotic medications are offset by serious negative medical consequences, including weight gain, obesity-related cardiovascular risk, insulin resistance, and diabetes. Behavioral interventions that aim to help people coping with serious mental illness to reduce weight, sustain weight loss, and achieve better fitness may improve the risk/benefit ratio of atypical antipsychotic medications. A small-group cognitive behavioral intervention that provides peer and structural risk-reduction support may be the most beneficial means of promoting healthy eating and exercise habits in people with serious mental illness who are living in group homes. This study will evaluate the effectiveness of a small-group cognitive behavioral intervention conducted in group homes for reducing significant medical risk factors often associated with people who have a serious mental illness and are taking atypical antipsychotic medications.

Participation in this study will last about 18 months through follow-up. All participants will undergo baseline assessments that will include the following: measurements of diet and exercise patterns, using self-report and observational methods; measurements of weight, body mass index, body fat distribution, pulse rate, and blood pressure; blood draws; and questions about psychological well-being and quality of life. Group homes will then be assigned randomly to provide participating residents with either the cognitive behavioral intervention or the time-matched attention control program. Participants in both groups will receive 26 weekly 1-hour small-group sessions and 26 weekly 30-minute individual sessions with a study facilitator. The cognitive behavioral sessions will focus on promoting healthy behaviors, dieting, and exercise. The time-matched attention control sessions will focus on improving communications, developing healthy techniques for coping with stress, and resolving conflicts. After completing treatment, all participants will receive 6 monthly 1-hour booster sessions of their assigned treatments. They will also repeat the baseline assessments 3 times over the following 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Resides in one of the designated group homes

Exclusion Criteria:

* Sufficiently impaired because of a psychiatric illness, as reflected in mental status in which informed judgment about study participation cannot be assured at the time of study entry
* Medical contraindication to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2006-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Average weight loss; body mass index; and effects across other behavioral, clinical, physiological, and ancillary measures | Measured at Month 12

SECONDARY OUTCOMES:
Ability of behavioral intervention to offset significant medical risk factors often associated with people living with mental illness | Measured at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Kelly, PhD, Principal Investigator — Medical College of Wisconsin; Carol L. Galletly, JD, PhD, Study Director — Medical College of Wisconsin; Anton M. Somlai, EdD, Study Director — Medical College of Wisconsin; Jill T. Owczarzak, PhD, Study Director — Medical College of Wisconsin; Timothy L. McAuliffe, PhD, Study Director — Medical College of Wisconsin; David W. Seal, PhD, Study Director — Medical College of Wisconsin; Thomas W. Heinrich, MD, Study Director — Medical College of Wisconsin